CLINICAL TRIAL: NCT02300805
Title: Accuracy of Endometrial Volume Measured by Virtual Organ Computer-aided AnaLysis (VOCAL)Versus Office Hysteroscopy for Diagnosis of Endometrial Polyps
Brief Title: Accuracy of Endometrial Volume Measured by VOCAL Versus Office Hysteroscopy for Diagnosis of Endometrial Polyps
Acronym: VOCAL
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, dr mohamed laban, professor mohammed laban, Ain Shams University
Other Study IDs: lab7681
Record Dates: First submitted 2014-11-18; First posted 2014-11-25 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Premenopausal; Metrorrhagia
Keywords: Endometrial volume , VOCAL , Endometrial , Metrorrhagia
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Endometrial volume will be assessed by 3DUS and VOCAL and compared to the results of office hysterscopy to measure the abilty of this technique to diagnose endometrial polyps in women complaining of abnormal uterine bleeding.

The safety of both procedures will be compared .

ELIGIBILITY:
Inclusion Criteria:

* Age more than 20 years
* Patients with irregular vaginal bleeding

Exclusion Criteria:

* Age less than 20 years
* Postmenopausal women
* presence of uterine fibroids
* Causes of vaginal bleeding due to systemic pathology , anticoagulant use , patients on hormonal contraception or using Intra Uterine Contraceptive Device ( IUCD ) .

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Premenopausal women complaining of irregular vaginal bleeding
Sampling Method: Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To measure the Safety and Tolerability" and "Efficacy of 3DUS versus office Hysteroscopy for diagnosis of endometrial polyps in premenopausal women | one year
  A prospective Observational Study

SECONDARY OUTCOMES:
To measure the best cut off value for endometrial volume (CC ) using Three Dimensional Sonography ( 3DUS and (VOCAL ) to diagnose endometrial polyps in women with premenopausal bleeding | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt